CLINICAL TRIAL: NCT05669794
Title: Real-world Effectiveness and Use of UPaDAcitinib in Patients With moderaTE-to-severe Atopic Dermatitis
Brief Title: An Observational Study to Assess Change in Disease Activity and Use of Upadacitinib Tablets in Adolescent and Adult Participants With Moderate to Severe Atopic Dermatitis in Real World
Acronym: UPDATE
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-628
Record Dates: First submitted 2022-12-21; First posted 2023-01-03 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; AD; Upadacitinib; RINVOQ
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Upadacitinib: Participants will receive upadacitinib as prescribed by their physician according to local label.

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. This study will assess how effective upadacitinib is in treating AD.

Upadacitinib is an approved drug for treating AD. Approximately 300 adolescent and adult participants who are prescribed upadacitinib by their physician in accordance with local label will be enrolled in France.

Participants will receive upadacitinib as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed up for approximately 24 months per participant and 30 days after last treatment dose for safety data collection.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Physician confirmed diagnosis of atopic dermatitis or atopic eczema at baseline.
* Symptom onset ≥1 year prior to baseline.
* Initiation of upadacitinib treatment for AD is indicated and prescribed per local label.
* The decision to prescribe upadacitinib is made prior to and independently of study participation.
* Participants who can understand and who are willing and able to complete the questionnaires, with parental support as required for adolescents.
* Participants (or legal representatives for adolescents) with a smartphone/tablet with internet access and willing to download the dedicated application to complete the questionnaires via this application.
* Participants (and legal representatives for adolescents) who have been informed verbally and in writing about this study before inclusion, and who do not object to their data being processed.
* Participants (and legal representatives for adolescents) able to understand and communicate with the investigator.

Exclusion Criteria:

* Participation in a clinical trial assessing an investigational drug, concurrently or within the last 30 days.
* Prior treatment with upadacitinib.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adolescent and adult participants with Atopic dermatitis (AD)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-02-21 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants achieving an absolute SCORing Atopic Dermatitis (SCORAD) of <25 | Month 4
  SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (59):
- France (59):
  - Ch Saint Quentin /Id# 249270, Saint-Quentin, Aisne
  - CHU Clermont-Ferrand /ID# 248611, Clermont, Auvergne-Rhône-Alpes
  - Hôpital Européen Marseille /ID# 257643, Marseille, Bouches-du-Rhone
  - Hopital Saint Joseph /ID# 255537, Marseille, Bouches-du-Rhone
  - Hopital Ponchaillou /ID# 251225, Rennes, Brittany Region
  - CHU Dijon /ID# 248984, Dijon, Cote-d Or
  - CH Georges Renon /ID# 248976, Niort, Deux-Sevres
  - CHU de Besancon - Jean Minjoz /ID# 248642, Besançon, Doubs
  - Hopitaux Drome Nord /ID# 248207, Romans-sur-Isère, Drome
  - CH Valence /ID# 250693, Valence, Drome
  - Centre Hospitalier de Quimper /ID# 251119, Quimper, Finistere
  - CHU Montpellier - Hopital Saint Eloi /ID# 251877, Montpellier, Herault
  - CHU nord - hopital Felix Guyon /ID# 250694, Saint-Denis, Le Reunion
  - Centre Hospitalier Saint-Nazaire /ID# 251200, Saint-Nazaire, Loire-Atlantique
  - Polyclinique Courlancy /ID# 250476, Reims, Marne
  - Hopital du Scorff /ID# 251226, Lorient, Morbihan
  - CHR Metz-Thionville - Hopital Bel-Air /ID# 252267, Thionville, Moselle
  - Centre Hospitalier de Valenciennes /ID# 258642, Valenciennes, Nord
  - Hopitaux Universitaires Henri Mondor - Hopital Henri Mondor /ID# 247209, Créteil, Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin /ID# 250807, Paris, Paris
  - CHU de Nantes, Hotel Dieu -HME /ID# 262563, Nantes, Pays de la Loire Region
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord /ID# 251117, St-Priest-en-Jarez, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 248864, Pierre-Bénite, Rhone
  - Centre Hospitalier du Mans /ID# 250510, Le Mans, Sarthe
  - Centre Hospitalier Métropole Savoie - Site Hôpital de Chambéry /ID# 252012, Chambéry, Savoie
  - CH Pontoise - Hopital René Dubos /ID# 248843, Pontoise, Val-d Oise
  - CH Avignon /ID# 251198, Avignon, Vaucluse
  - CHI POISSY - Saint-Germain-en-Laye /ID# 248612, Saint-Germain-en-Laye, Yvelines
  - Hopital Nord Amiens /ID# 250300, Amiens
  - Chu Angers /Id# 248674, Angers
  - CH Victor Dupouy /ID# 247216, Argenteuil
  - Centre Hospitalier de Béziers /ID# 264454, Béziers
  - Hopital Ambroise Pare /ID# 253337, Boulogne-Billancourt
  - CHU de CAEN - Hopital de la Cote de Nacre /ID# 252127, Caen
  - CH de Cahors /ID# 251190, Cahors
  - Centre Hospitalier de Calais /ID# 249449, Calais
  - Cabinet Dermatologie et Esthetique /ID# 247972, Cannes
  - CH William Morey /ID# 256417, Chalon-sur-Saône
  - CH Annecy Genevois - Site Annecy /ID# 249024, Epagny Metz Tessy
  - CH la Rochelle /ID# 252128, La Rochelle
  - CH Emile Roux Le Puy en Velay /ID# 248983, Le Puy-en-Velay
  - Hopital Saint Vincent de Paul /ID# 247218, Lille
  - CHU Limoges - Dupuytren 2 /ID# 251224, Limoges
  - Hopital Femme Mere Enfant /ID# 258682, Lyon
  - Cideazur /ID# 247905, Nice
  - Hôpital Saint-Louis /ID# 251228, Paris
  - Cabinet libéral du Dr KURIHARA /ID# 249664, Paris
  - Hopital Bichat-Claude Bernard /ID# 251274, Paris
  - CH de PAU /ID# 248567, Pau
  - Hôpital Charles-Nicolle /ID# 247215, Rouen
  - CHU de Rouen /ID# 250648, Rouen
  - Hôpital d'instruction des armées Bégin /ID# 247751, Saint-Mandé
  - Ch Salon de Provence /Id# 248829, Salon-de-Provence
  - Hôpital d'Instruction des Armées Sainte-Anne /ID# 247908, Toulon
  - CHU Toulouse - Hopital Larrey /ID# 247219, Toulouse
  - Hopital Nord Franche Comté /ID# 261628, Trévenans
  - Cabinet Liberal /ID# 251195, Villeurbanne
  - Hopital Prive d'Antony /ID# 247324, Antony, Île-de-France Region
  - Hopital Pitie Salpetriere /ID# 253464, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related info — https://www.abbvieclinicaltrials.com/study/?id=P23-628